CLINICAL TRIAL: NCT01971437
Title: A Randomised Study of Cystoscopy and Cystodistension Versus Cystoscopy Alone in Women With Overactive Bladder Syndrome.
Brief Title: Cystoscopy and Cystodistension; Therapeutic and Aetiological Aspect in Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Jonathan Duckett, Consultant Gynaecologist, Medway NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBC
Record Dates: First submitted 2013-10-21; First posted 2013-10-29 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Incontinence, Urge
Keywords: Overactive Bladder; OAB; Cystoscopy; Cystodistension; UTI; Cytokines
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Cystoscopy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cystodistension & Cystoscopy Arm (Experimental): This is the Arm receiving cystodistension and cystoscopy due to refractory OAB.
  Interventions: Procedure: Cystodistension & Cystoscopy
- Cystoscopy Arm (Placebo Comparator): This is the arm that receives cystoscopy only in women with refractory OAB.
  Interventions: Procedure: Cystodistension & Cystoscopy

INTERVENTIONS:
Procedure: Cystodistension & Cystoscopy — Women with refractory OAB receiving Cystoscopy and cystodistension
  Other Names: Cystodistension; Cystoscopy; OAB; Treatments

SUMMARY:
This is an ethically approved randomised controlled study looking at whether Cystodistension(filling the bladder with fluid under pressure) provides any benefit over cystoscopy alone (looking in the bladder) in women with refractory overactive bladder. Urine samples will also be assessed for underlying infected cause of OAB using urinalysis, microscopy and culture and cytokine assays (In collaboration with the University of Kent). We hypothesize that Cystodistension has a therapeutic benefit to women with refractory OAB and the there is an increase prevalence in chronic urinary infections with raised cytokines in women with refractory OAB.

DETAILED DESCRIPTION:
We aim to measure outcomes initially, 6 weels and 6months follow-up.

1. Resolution measured by Urgency Perception Scale (UPS). Resolution of urgency will be assessed with the UPS. The numbers of women with a Level 3 UPS score (hold and finish task) will be compared using Chi square test in patients treated with cystodistension vs non cystodistension arms.
2. Change in quality of life status determined by quality of life questionnaires will ismilarly be comapred between the 2 arms of the study.
3. Change in urinary symptoms defined by Patient's Perception of Intensity Scale. Change in uregncy scores will be compared between the 2 arms of the study.

Secondary Outcome Measure:1. Prevalence of chronic urinary infection and organisms in patients with refractory OAB 2. To identify whether urinary cytokines are present in a higher proportion of patients with OAB.

Inclusion Criteria

1. Women with only OAB symptoms
2. Women who have failed bladder drill and anticholinergic agents
3. Women who stopped medication due to side-effects or lack of efficacy
4. Currently receiving no treatment

Exclusion Criteria

1. Patient with co-existing urodynamic stress incontinence
2. Patients with neurological diseases
3. Patients with pre-existing voiding dysfunction

ELIGIBILITY:
Inclusion Criteria

1. Women with only OAB symptoms
2. Women who have failed bladder drill and anticholinergic agents
3. Women who stopped medication due to side-effects or lack of efficacy
4. Currently receiving no treatment

Exclusion Criteria

1. Patients with co-existing urodynamic stress incontinence
2. Patients with neurological diseases
3. Patients with pre-existing voiding dysfunction

   * Free flow rate <5th centile or equivalent reduced pressure flow rate OR
   * Post-void residual volume greater than 100ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess the presence of urgency and urge incontinence initially, 6 weeks and 6 months | 12-18months
  1. Resolution measured by Urgency Perception Scale.
  2. Change in quality of life status.
  3. Change in urinary symptoms defined by the Patient's Perception of Intensity Scale

SECONDARY OUTCOMES:
Improved quality of life. | 12-18 months
  Change in quality of life status, Urgency Perception Scale and Patient's Perception of Intensity Scale scoring initially, 6 weeks and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan RA Duckett, FRCOG, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway Maritime Hospital, Gillingham, Kent, United Kingdom